CLINICAL TRIAL: NCT00537511
Title: A Multicenter, Phase I/IIA, Open-Label, Dose-Escalation Study to Determine the Maximum Tolerated Dose and To Evaluate the Safety Profile of CC-4047 Administered in Combination With Cisplatin and Etoposide in Patients With Extensive Disease Small Cell Lung Cancer
Brief Title: A Phase I/II Study to Determine the Maximum Tolerated Dose (MTD) and Safety of CC-4047 (Pomalidomide) Administered in Conjunction With Cisplatin and Etoposide
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated for administrative reasons.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-SCLC-002
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Small Cell
MeSH Terms: conditions — Carcinoma, Small Cell | interventions — pomalidomide; Cisplatin; Etoposide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose-finding arm: Pomalidomide + Cisplatin + Etoposide (Experimental): Oral pomalidomide 1 mg - 5 mg daily (QD) for 14 consecutive days of a 21-day cycle, in combination with intravenous (IV) cisplatin 25 mg/m^2 and IV etoposide 100 mg/m^2 on Days 1, 2 and 3 of each cycle during the dose-finding phase (Treatment and Extension Periods; 6 cycles in total). Dose escalation followed a standard phase 1 3+3 design. Participants continuing took only their pomalidomide dose (monotherapy) for an additional 3-week Recovery Period (14 days of consecutive dosing followed by 7 days of no study medication). Participants continuing took oral pomalidomide 5 mg QD as monotherapy for 14 consecutive days of each 21-day cycle until disease progression in the Maintenance Phase.
  Interventions: Drug: Pomalidomide; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Pomalidomide
  Other Names: CC-4047; Pomalyst
Drug: Cisplatin
  Other Names: Cisplatinum; CDDP; Platin
Drug: Etoposide
  Other Names: Etoposide phosphate; VP-16; Etopophos

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and safety of CC-4047 (pomalidomide) given in combination with cisplatin and etoposide in patients with extensive disease small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* signature of informed consent
* Age >= 18
* histologically or cytologically confirmed small cell lung cancer (SCLC)
* extensive stage SCLC
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2
* brain metastases that are asymptomatic and do not require steroid control
* females of child bearing potential must use two forms of birth control

Exclusion Criteria:

* pregnant or lactating females
* prior use of cytotoxic chemotherapy
* surgery within 14 days of study
* radiation within 14 days of study
* prior therapy with CC-4047 (pomalidomide), lenalidomide or thalidomide
* concurrent use or anticipated use of anti-cancer agents
* absolute neutrophil count (ANC) < 1500/mm^3
* platelets < 100 x 10^3/µL
* serum creatinine >2.5 mg/dL
* serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) > 3.0 x upper limit of normal (ULN)
* serum total bilirubin > 1.8 mg/dL
* uncontrolled hypercalcemia
* creatinine clearance <50 mL/min
* uncontrolled hypertension
* neuropathy >= grade 2
* body mass index (BMI) >= 40
* any other active invasive malignancy requiring treatment
* known chronic infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)
* inability or unwillingness to comply with birth control requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2010-11-01 (Actual); Study Completion 2010-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Jungnelius, MD, Study Director — Celgene Corporation
Locations (6):
- United States (3):
  - Ireland Cancer Center, Case Western Reserve University, Division of Hematology/Oncology, Cleveland, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Canada (3):
  - Juranvinski Cancer Center - Medical Oncology, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Mc Gill University - Department of Oncology - Clinical Research Program, Montreal, Quebec

REFERENCES:
- [Result] Ellis PM, Jungnelius U, Zhang J, Fandi A, Beck R, Shepherd FA. A phase I study of pomalidomide (CC-4047) in combination with cisplatin and etoposide in patients with extensive-stage small-cell lung cancer. J Thorac Oncol. 2013 Apr;8(4):423-8. doi: 10.1097/JTO.0b013e318282707b. PMID 23370364

RESULTS

PARTICIPANT FLOW:
Groups:
- Pomalidomide (Overall): Oral pomalidomide 1 mg - 5 mg daily (QD) for 14 consecutive days of a 21-day cycle, in combination with intravenous (IV) cisplatin 25 mg/m^2 and IV etoposide 100 mg/m^2 on Days 1, 2 and 3 of each cycle during the dose-finding phase (Treatment and Extension Periods; 6 cycles in total). Dose escalation followed a standard phase 1 3+3 design. Participants continuing took only their pomalidomide dose (monotherapy) for an additional 3-week Recovery Period (14 days of consecutive dosing followed by 7 days of no study medication). Participants continuing took oral pomalidomide 5 mg QD as monotherapy for 14 consecutive days of each 21-day cycle until disease progression in the Maintenance Phase.
Period: Treatment Period (Combination)
Arm/Group | Pomalidomide (Overall)
Started | 22
Intent-to-Treat (ITT) Populaton | 22 (ITT = all participants enrolled in the study.)
Safety Population | 22 (Safety = All participants who took ≥1 dose of study treatment.)
Completed | 17
Not Completed | 5
Period: Extension Period (Combination)
Arm/Group | Pomalidomide (Overall)
Started | 17
Completed | 11
Not Completed | 6
Period: Recovery Period (Monotherapy)
Arm/Group | Pomalidomide (Overall)
Started | 11
Completed | 3
Not Completed | 8
Period: Maintenance Phase (Monotherapy)
Arm/Group | Pomalidomide (Overall)
Started | 8
Completed | 0
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | Pomalidomide (Overall)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White) | 22
  Non-caucasian | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose level at which no more than 1 in 6 participants experienced a dose-limiting toxicity (DLT) during the first 21-day cycle of treatment. The MTD Phase included the Treatment period (Cycle 1: Identification of the MTD) and the Extension period (Cycles 2 to 6: Confirmation of Safety of the MTD). (See Secondary Outcome Measure 2 for data on DLTs.)
Time Frame: Cycle 1 (21 days)
Population: Safety Population
Measure: Number; unit: mg
Arm/Group | Pomalidomide (Overall)
Number analyzed (Participants) | 22
mg | 4

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) During the MTD Phase
Description: For the purposes of determining the MTD (see Primary Outcome Measure), a DLT was defined as any 1 or more of the following: inability to deliver all 3 doses of cisplatin and etoposide due to toxicity; inability to deliver 14 consecutive days of daily pomalidomide dosing because the participant did not tolerate the medication due to any of the following: ≥ grade 3 non-hematological toxicity (excluding alopecia) occurring before Day 14 of pomalidomide dosing; febrile neutropenia (absolute neutrophil count [ANC] <1,000/µL and fever >101ºF, core temperature); grade 4 neutropenia of ≥7 days duration with onset on or before Day 14 of pomalidomide dosing; platelet count <25,000/µL occurring before Day 14 of pomalidomide dosing. National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), Version 4.0, grades: 1=mild, 2=moderate, 3=severe, 4=life threatening, 5=death.
Time Frame: Cycles 1 - 6 (21-day cycles)
Population: Safety Population
Measure: Number; unit: participants
Groups:
- Pomalidomide 1 mg: Oral pomalidomide 1 mg QD for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
- Pomalidomide 3 mg: Oral pomalidomide 3 mg QD for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
- Pomalidomide 4 mg: Oral pomalidomide 4 mg QD for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
- Pomalidomide 5 mg: Oral pomalidomide 5 mg QD for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
Arm/Group | Pomalidomide 1 mg | Pomalidomide 3 mg | Pomalidomide 4 mg | Pomalidomide 5 mg
Number analyzed (Participants) | 6 | 4 | 6 | 6
participants | 1 | 0 | 0 | 2

3. Secondary Outcome: Tumor Response Rate According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Investigator's best assessment of response based on RECIST criteria during the MTD phase. For target lesions: Complete Response (CR)=Disappearance of all target lesions; Partial Response (PR)=≥30% decrease in sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD; Progressed Disease (PD)=≥20% increase in sum of LD of target lesions taking as reference the smallest sum LD recorded since treatment started or the appearance of ≥1 new lesions; Stable Disease (SD)=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum LD since treatment started. For non-target lesions: CR= Disappearance of all non-target lesions and normalization of tumor marker level; Incomplete Response/SD=Persistence of ≥1 non-target lesions and/or maintenance of tumor marker level above normal limits; PD=Appearance of ≥1 new lesions; unequivocal progression of existing non-target lesions.
Time Frame: Cycles 1 -6 (21-day cycles)
Population: ITT population. 'Not Assessed' category includes participants who did not have adequate data for response assessment at baseline and/or post-baseline prior to the use of any non-protocol anti-tumor therapy.
Measure: Number; unit: participants
Groups:
- Pomalidomide (Overall, MTD Phase): Participants received daily oral pomalidomide 1 mg to 5 mg for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
Arm/Group | Pomalidomide 1 mg | Pomalidomide 3 mg | Pomalidomide 4 mg | Pomalidomide 5 mg | Pomalidomide (Overall, MTD Phase)
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 22
participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 3 | 3 | 2 | 3 | 11
  No Change/Stable Disease | 0 | 0 | 0 | 0 | 0
  Progressive Disease | 1 | 1 | 1 | 1 | 4
  Not Assessed | 0 | 0 | 1 | 0 | 1
  Missing | 2 | 0 | 2 | 2 | 6

4. Secondary Outcome: Duration of Response
Description: Duration of Response was calculated from first Partial Response (PR) or Complete Response (CR) to disease progression. Duration of response was censored at the last date that the participant was known to be progression-free for: 1) participants who had not progressed at the time of analysis; 2) participants who had been removed from the treatment phase prior to documentation of progression.
Time Frame: From first Partial Response (PR) or Complete Response (CR) to disease progression (maximum of 19.4 weeks)
Population: Number of participants in ITT population who were considered Responders.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Pomalidomide (Overall)
Number analyzed (Participants) | 11
weeks | 13.2 (5.54)

5. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as time (in weeks) from enrollment to death. The median is based on Kaplan-Meier estimate, with 95% confidence intervals about the median overall survival. Overall survival was censored at the last time participant was known to be alive for those who were alive at time of analysis.
Time Frame: From enrollment through study termination (approximately 35 months)
Population: Participants in the ITT population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pomalidomide (Overall)
Number analyzed (Participants) | 22
weeks | 49.6 [28.0 to 63.9]

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the MTD (Combination Treatment) Phase
Description: Adverse event (AE) = any noxious, unintended, or untoward medical occurrence occurring at any dose that may appear or worsen in a participant during the course of a study, including new intercurrent illness, worsening concomitant illness, injury, or any concomitant impairment of participant's health, including laboratory test values, regardless of etiology. Serious adverse event (SAE) = any AE which: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. TEAE = any AE occurring or worsening on or after the first treatment with any study drug. Related = suspected by investigator to be related to study treatment. National Cancer Institute [NCI] Common Toxicity Criteria for Adverse Events [CTCAE], Version 4.0, grades: 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, 5 = death.
Time Frame: Cycles 1-6 (21-day cycles). Median (full range) duration of exposure (in weeks) to pomalidomide (MTD Phase): 1 mg, 17.9 (1.0, 20.3); 3 mg, 17.0 (16.9, 22.0); 4 mg, 14.0 (0.7, 22.0); 5 mg, 13.0 (2.0, 22.1). Cisplatin and etoposide: 15.3 (0.4, 20.6).
Population: Safety population
Measure: Number; unit: participants
Groups:
- Pomalidomide 1 mg: Participants received daily oral pomalidomide 1 mg for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
- Pomalidomide 3 mg: Participants received daily oral pomalidomide 3 mg for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
- Pomalidomide 4 mg: Participants received daily oral pomalidomide 4 mg for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
- Pomalidomide 5 mg: Participants received daily oral pomalidomide 5 mg for 14 consecutive days of a 21-day cycle in combination with cisplatin 25 mg/m^2 and etoposide 100 mg/m^2 administered intravenously (IV) on Days 1, 2 and 3 of each cycle during the MTD Phase (6 cycles in total).
Arm/Group | Pomalidomide 1 mg | Pomalidomide 3 mg | Pomalidomide 4 mg | Pomalidomide 5 mg | Pomalidomide (Overall, MTD Phase)
Number analyzed (Participants) | 6 | 4 | 6 | 6 | 22
participants
  ≥1 TEAE | 6 | 4 | 6 | 6 | 22
  ≥1 TEAE related to pomalidomide (POM) | 6 | 4 | 6 | 6 | 22
  ≥1 TEAE related to cisplatin and/or etoposide(C/E) | 6 | 4 | 6 | 6 | 22
  ≥1 Grade 3 or higher (GR3+) TEAE | 6 | 4 | 6 | 6 | 22
  ≥1 GR 3+ TEAE related to POM | 3 | 2 | 4 | 5 | 14
  ≥1 GR 3+ TEAE related to C/E | 6 | 3 | 6 | 5 | 20
  ≥1 Serious TEAE | 3 | 1 | 3 | 3 | 10
  ≥1 Serious TEAE related to POM | 2 | 1 | 1 | 3 | 7
  ≥1 Serious TEAE related to C/E | 2 | 1 | 3 | 3 | 9
  ≥1 TEAE leading to (→) withdrawal of POM | 2 | 0 | 2 | 2 | 6
  ≥1 TEAE → withdrawal of C/E | 2 | 1 | 1 | 2 | 6
  ≥1 TEAE → dose reduction/interruption of POM | 5 | 2 | 4 | 4 | 15
  ≥1 TEAE → dose reduction/interruption of C/E | 3 | 3 | 3 | 4 | 13

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the Recovery Period or Maintenance (Monotherapy) Phase
Description: Adverse event (AE) = any noxious, unintended, or untoward medical occurrence occurring at any dose that may appear or worsen in a participant during the course of a study, including new intercurrent illness, worsening concomitant illness, injury, or any concomitant impairment of participant's health, including laboratory test values, regardless of etiology. TEAE = any AE occurring or worsening on or after the first treatment with any study drug. 'Related' = suspected by investigator to be related to study treatment. National Cancer Institute [NCI] Common Toxicity Criteria for Adverse Events [CTCAE], Version 4.0, grades: 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, 5 = death.
Time Frame: Cycle 7 to discontinuation (21-day cycles). Median (full range) duration of exposure (in weeks) to pomalidomide during Maintenance Phase was 5.0 (1.1, 36.0).
Population: Safety population; participants continuing in the Recovery Period and Maintenance Phase.
Measure: Number; unit: participants
Arm/Group | Pomalidomide (Overall)
Number analyzed (Participants) | 11
participants
  ≥1 TEAE | 9
  ≥1 TEAE related to pomalidomide (POM) | 8
  ≥1 TEAE related to cisplatin and/or etoposide (C/E | 7
  ≥1 Grade 3 or higher (GR3+) TEAE | 6
  ≥1 GR 3+ TEAE related to POM | 2
  ≥1 GR 3+ TEAE related to C/E | 2
  ≥1 TEAE → dose reduction/interruption of POM | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were defined as any AE occurring or worsening on or after the first treatment of the study medication and within 30 days after the last dose. See Additional Description for duration of exposure for each treatment.
Description: Median (full range) duration of exposure (in weeks) to pomalidomide (MTD Phase): 1 mg, 17.9 (1.0, 20.3); 3 mg, 17.0 (16.9, 22.0); 4 mg, 14.0 (0.7, 22.0); 5 mg, 13.0 (2.0, 22.1). Cisplatin and etoposide: 15.3 (0.4, 20.6). Pomalidomide (Maintenance Phase): 5.0 (1.1, 36.0).
Arm/Group | Pomalidomide 1 mg | Pomalidomide 3 mg | Pomalidomide 4 mg | Pomalidomide 5 mg | Pomalidomide (Overall)
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/4 | 3/6 | 3/6 | 10/22
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 6/6 | 6/6 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide 1 mg (N=6) | Pomalidomide 3 mg (N=4) | Pomalidomide 4 mg (N=6) | Pomalidomide 5 mg (N=6) | Pomalidomide (Overall) (N=22)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 2
Atrioventricular Block Complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Diverticular Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1
Neutropenic Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide 1 mg (N=6) | Pomalidomide 3 mg (N=4) | Pomalidomide 4 mg (N=6) | Pomalidomide 5 mg (N=6) | Pomalidomide (Overall) (N=22)
Fatigue (General disorders) | 5 | 4 | 6 | 6 | 21
Oedema peripheral (General disorders) | 2 | 1 | 3 | 3 | 9
Asthenia (General disorders) | 1 | 1 | 0 | 1 | 3
Chest discomfort (General disorders) | 1 | 0 | 1 | 1 | 3
Chest pain (General disorders) | 0 | 0 | 2 | 1 | 3
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 3
Chills (General disorders) | 0 | 0 | 1 | 1 | 2
Irritability (General disorders) | 1 | 0 | 0 | 1 | 2
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 1
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 1
Infusion site reaction (General disorders) | 0 | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 5 | 5 | 15
Constipation (Gastrointestinal disorders) | 3 | 2 | 4 | 4 | 13
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 1 | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 6
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 2 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 3 | 2 | 2 | 9
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 2 | 6
Dysgeusia (Nervous system disorders) | 2 | 2 | 2 | 0 | 6
Headache (Nervous system disorders) | 0 | 0 | 4 | 0 | 4
Tremor (Nervous system disorders) | 2 | 0 | 1 | 0 | 3
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 5 | 12
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 4 | 0 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 3 | 5 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 2 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 2 | 2 | 2 | 3 | 9
Weight decreased (Investigations) | 0 | 2 | 0 | 1 | 3
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1 | 2
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Electrocardiogram qt prolonged (Investigations) | 0 | 1 | 0 | 0 | 1
Electrocardiogram st-t segment abnormal (Investigations) | 1 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 3 | 5
Flushing (Vascular disorders) | 1 | 1 | 0 | 1 | 3
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 1 | 1 | 4
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Lacrimation increased (Eye disorders) | 1 | 1 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 2
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 2 | 3
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 1 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 2
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 2
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon investigator submission of a publication or presentation to Celgene, Celgene shall complete its review within 60 days after receipt of the proposed publication or presentation. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of property of Celgene that would be affected by such proposed publication or presentation.